CLINICAL TRIAL: NCT06617468
Title: Effect of the Computer Aided Diagnosis with Explainable Artificial Intelligence for Colon Polyp on Optical Diagnosis and Acceptance of Technology
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Su Jin Chung, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2311-049-1482
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Colon Polyp
Keywords: colon polyp; optical diagnosis; computer-aided diagnosis
MeSH Terms: conditions — Colonic Polyps | interventions — Diagnosis, Computer-Assisted; Deep Learning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- computer-aided diagnosis with explainable AI (Experimental): Perform a same test to estimate the pathologic diagnosis on 200 NBI still images with computer-aided diagnosis with explainable AI
  Interventions: Diagnostic Test: computer-aided diagnosis with explainable AI
- computer-aided diagnosis with deep learning (Active Comparator): Perform a same test to estimate the pathologic diagnosis on 200 NBI still images with computer-aided diagnosis with deep learning
  Interventions: Diagnostic Test: computer-aided diagnosis with deep learning

INTERVENTIONS:
Diagnostic Test: computer-aided diagnosis with explainable AI — Perform a same test to estimate the pathologic diagnosis on 200 NBI still images with computer-aided diagnosis with explainable AI.
  Arms: computer-aided diagnosis with explainable AI
Diagnostic Test: computer-aided diagnosis with deep learning — Perform a same test to estimate the pathologic diagnosis on 200 NBI still images with computer-aided diagnosis with deep Iearning.
  Arms: computer-aided diagnosis with deep learning

SUMMARY:
The goal of this clinical trial is to learn if computer-aided diagnosis with deep learning and computer-aided diagnosis with explainable AI work to optical diagnosis performance and acceptance of technology in endoscopists. The main questions it aims to answer are:

Do computer-aided diagnosis with deep learning and computer-aided diagnosis with explainable AI improve optical diagnosis performance in endoscopists?

Does experience using deep learning-based computer-assisted diagnosis and explainable AI-based computer-assisted diagnosis improve endoscopists' acceptance of computer-aided diagnosis as a technology?

Participants will:

Conduct a survey on acceptance and use of technology about computer-aided diagnosis.

Perform a test to estimate the pathologic diagnosis on 200 NBI still images without the aid of computer-aided diagnosis.

More than 1 month later, perform a same test to estimate the pathologic diagnosis on 200 NBI still images with computer-aided diagnosis with deep learning or explainable AI.

Conduct a survey on acceptance and use of technology about computer-aided diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopists with colonoscopy experience

Exclusion Criteria:

* Who can not perform colonoscopy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of optical diagnosis | From baseline test to the follow up test (more than 1 month later from baseline test)
  The proportion of cases in which pathological results are consistent with endoscopic estimation of adenoma and hyperplastic polyp

SECONDARY OUTCOMES:
acceptance of computer-aided diagnosis as a technology | From baseline test to the follow up test (more than 1 month later from baseline test)
  Survey on acceptance and use of technology about computer-aided diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Healthcare System Gangnam Center, Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No